CLINICAL TRIAL: NCT03233334
Title: Purpose Project: Reclaiming Life Purpose After Breast Cancer (Feasibility Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Mary Radomski, Senior Scientific Advisor, Allina Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CKMR-1702
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Purpose Project Group (Experimental): Group receiving Purpose Project intervention.
  Interventions: Behavioral: Purpose Project

INTERVENTIONS:
Behavioral: Purpose Project — The purpose project intervention 8-session group intervention that integrates education, support, self-reflection, and action-expectation to help people reaffirm or reconstruct self-grounded purpose after significant life events/transitions. The 8 sessions extend over 2-3 months, with 7 weekly sessions and the final session 1 month after Session 7. The intervention is structured around the 6 dimensions of flourishing (autonomy, self-acceptance, personal growth, relationships, purpose in life, external mastery), the goal of which is to help people enact behaviors that move them forward in reframing a sense of self and reaffirming or reconstructing a sense of purpose in life that helps them flourish.

SUMMARY:
The Purpose Project intervention is an 8-session progressive structure that was developed based on theoretical and scientific evidence from psychology and occupational therapy. The goal of the intervention is to provide participants with information, tools, and support that help them move towards reclaiming a sense of self-grounded purpose in daily life. The study will use a convenience sample of women with breast cancer to evaluate the feasibility of the Purpose Project intervention in terms of demand/acceptability, implementation, and limited-efficacy testing. Findings will be used to inform a later study to evaluate the efficacy of the Purpose Project intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Between 25 and 74 years of age
2. Completed chemotherapy and/or radiation treatment for Stage 1, 2, or 3 breast cancer up to 5 years prior to study enrollment
3. English speaking
4. Graduated from high school
5. Able to see, hear, speak (with or without assistive devices)
6. Able to provide own transportation to sessions
7. Willing and able to commit to attend all 8 intervention sessions, 2 testing sessions, and the one-to-one interview that occurs after completing the 8 intervention sessions.

Exclusion Criteria:

1. Stage 4 breast cancer or any other stage 4 cancer
2. Actively receiving chemotherapy or radiation treatments for cancer. (However, patients may be on Herceptin and/or endocrine treatment and participate in the study.)
3. History of neurologic disorder (such as stroke or brain injury) with residual impairments that likely interfere with learning
4. Any medical condition (physical or mental health) that interferes with the performance of everyday activities and roles.

Ages: 25 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change in psychological well-being | Will be administered at Week 0 (pre-testing) and at Week 12 (session 8).
  Using the Psychological Scales of Wellbeing questionnaire (Ryff, 1989; Ryff, & Keyes, 1995), psychological wellbeing pre- and post- intervention will be tracked.

SECONDARY OUTCOMES:
Recruitment | Up to 1 month after IRB approval
  Number of prospective participants approached by clinicians and number of self-referred prospective participants who contact PI or Study Coordinator with inquiries about the study
Time of pre-testing session | Duration of pre-testing session (approximately 2 hours) at week 0 to week 1
  Actual length (in minutes) of pre-testing session.
Time of testing session | Each week from week 2 through week 8, approximately 2.5 hours at each session
  Actual length (in minutes) of testing session.
Time of post-testing session | Duration of session 8 (at week 12), approximately 2 hours
  Actual length (in minutes) of testing session.
Homework completion | Each week from week 2 through week 8
  Whether or not homework was attempted
Intervention fidelity | Each week from week 2 through week 8
  Which key intervention elements were provided during a given session
Change in Meaning in life | At week 0 and at week 12
  Meaning in Life Questionnaire (Steger et al., 2006): A 10-item questionnaire designed to measure 2 dimensions of meaning in life: Presence of Meaning (how much respondents feel their lives have meaning) and Search for Meaning (how much respondents strive to find meaning and understanding in their lives).
Change in Satisfaction with Participation in Discretionary Social Activities | At week 0 and at week 12
  Satisfaction with Participation in Discretionary Social Activities (Hahn et al., 2010): Self-report questionnaires in which participants rated their level of satisfaction (1-5 scale) with social roles (14 items) and discretionary activities (12 items).
Engagement in Meaningful Activities | At week 0 and at week 12
  Engagement in Meaningful Activities Survey (Eakman, 2010):A 12-item self-report questionnaire designed to measure the extent to which a person experiences meaningfulness in his/her daily life activities.
Purpose Status and Expectations | At Week 12
  A 2-question self-report developed by the study team to better understand what participants' hope to gain during the study and perceived changes.
Participant Experience of Purpose Project | At week 12 and at week 14-20
  Participant experience of purpose project as measured by self-report questionnaire and post-intervention interview.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Radomski, PhD, OTR/L, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No